CLINICAL TRIAL: NCT02131753
Title: Therapy Optimisation for the Treatment of Hairy Cell Leukemia
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Giessen (Other)
Responsible Party: Principal Investigator, Jurgen Barth, Head of StiL Coordinating Center, University of Giessen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NHL 3-2004
Record Dates: First submitted 2014-04-30; First posted 2014-05-06 (Estimated); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Hairy Cell Leukemia
Keywords: hairy cell leukemia; untreated; cladribine subcutaneous
MeSH Terms: conditions — Leukemia, Hairy Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cladribine s.c. injection, HCL treatment (Other): Cladribine 0.14 mg/kg body weight for 5 consecutive days (d 1 - 5) as subcutaneous bolus injection for patients with hairy cell leukemia needing treatment
  Interventions: Drug: Cladribine s.c. injection, HCL treatment

INTERVENTIONS:
Drug: Cladribine s.c. injection, HCL treatment — Patients with hairy cell leukemia and the need for treatment are given cladribine 0.14 mg/kg for 5 consecutive days as a s. c bolus injection
  Other Names: Litak(R); 2-CdA

SUMMARY:
The trial will test the effectiveness and toxicity of subcutaneous treatment with one cycle of cladribine in patients with hairy cell leukemia requiring treatment.

They have to be untreated so far or may be pretreated with alpha-interferon.

DETAILED DESCRIPTION:
Evaluation of remission status will take place 4 months after treatment. In addition, it will be tested whether patients with non-optimal response will have a benefit from a second cycle of cladribine.

Non-optimal response is: patients with detectable residual disease; achievement of partial remission or detectable residual infiltration in the bone marrow.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically verified hairy cell leukemia
* Presence of hairy cells in the bone marrow and peripheral blood detected by positive TRAP staining and / or co expression if cell surface antigens cluster of differentiation (CD) 19/CD25 or CD19/CD103 (b-ly7)
* No previous cytostatic treatment (splenectomy or interferon treatment are allowed)
* Need for treatment
* Age at least 18 years old
* General state of health according to WHO 0-2
* Current histology, not older than 6 months
* Written consent by patient

Exclusion Criteria:

* Patients not fulfilling inclusion criteria above
* Hairy cell leukemia variants (HCL-V): presence of lymphoid cells in bone marrow and / or peripheral blood, which have an intermediate morphology between hairy cells and prolymphocytes (negative TRAP staining and co- expression of CD19/CD103 without CD25
* Pretreatment with purine analogues or other chemotherapeutics
* Concomitant corticosteroid therapy
* Severe dysfunction of the heart (NYHA III or IV), the lung (WHO-Grade III or IV), the liver, except due to lymphoma (bilirubin > 2 mg/dl, alkaline phosphatase, glutamate-oxalacetate transaminase and glutamate-pyruvate transaminase > 2 x upper limit of normal), the kidneys (creatinin > 2 mg/dl or creatinine clearance < 50 ml/min), central nervous system diseases including psychoses.
* Proven HIV infection
* Active Hepatitis
* Other florid infections
* Anamnesis / diagnosis of other malignant disease (other than non-melanoma associated skin tumours or stage 0 in situ carcinoma of the cervix)
* Pregnant or lactating women

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2004-05; Primary Completion 2025-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Determination of the rate of complete remissions after one cycle with subcutaneous cladribine | 4 months after treatment

SECONDARY OUTCOMES:
Rate of complete remissions in patient who still have detectable residual disease | 4 months after treatment
  A second cycle of cladribine after an interval of 4 months following the first cycle.

OTHER OUTCOMES:
Overall effectiveness | 20 years
  Determination of:
  * overall remission rate
  * duration of remission
  * immunodeficiency induced by treatment, its duration, infectious and other complications resulting from that
  * frequency of secondary neoplasia during life long follow up
  * overall survival
Improvement of remission deepness | Date of staging after first cycle + 4 months
  Can a complete remission be achieved with a second cycle in patients who have achieved only a partial remission after one cycle?
Improvement of remission quality | Date of staging after first cycle + 4 months
  Can the quality of remission achieved with the first cycle be improved with a second cycle?
Lowering risk of relapse | Date of proven remission until the date of firdt documented progression or date of death from any cause, whichever came first, assessed up to 20 years
  Can the expected risk of relapse be lowered and the duration of remission be prolonged?

CONTACTS AND LOCATIONS:
Overall Officials: Mathias J Rummel, Prof. Dr., Principal Investigator — Justus-Liebig-University | University Hospital | Medicinal Clinic IV
Locations (74):
- Germany (74):
  - Community based hemato-oncology medical office, Ansbach
  - Community based hemato-oncology medical office, Aschaffenburg
  - Rhön-Saale-Klinik gGmbH, Bad Neustadt an der Saale
  - Community based hemato-oncology medical office, Berlin
  - Charité - Universitätsmedizin Berlin, Berlin
  - Community based hemato-oncology medical office, Bremen
  - Community based hemato-oncology medical office, Celle
  - Community based hemato-oncology medical office, Cottbus
  - Community based hemato-oncology medical office, Darmstadt
  - Community based hemato-oncology medical office, Dresden
  - Community based hemato-oncology medical office, Duisburg
  - Klinik Duisburg-West, Duisburg
  - Universitätsklinik Düsseldorf, Düsseldorf
  - Community based hemato-oncology medical office, Ehingen
  - Community based hemato-oncology medical office, Erlangen
  - Community based hemato-oncology medical office, Frankfurt
  - Krankenhaus Nordwest, Frankfurt
  - Community based hemato-oncology medical office, Freiburg im Breisgau
  - Community based hemato-oncology medical office, Friedrichshafen
  - Community based hemato-oncology medical office, Fürth
  - Community based hemato-oncology medical office, Germering
  - Community based hemato-oncology medical office, Giessen
  - University Clinic | Medicinal Clinic IV, Giessen
  - St.-Marien-Hospital, Hagen
  - Community based hemato-oncology medical office, Halle
  - Evangelisches Krankenhaus, Hamm
  - Community based hemato-oncology medical office, Hanau
  - Community based hemato-oncology medical office, Heidelberg
  - Community based hemato-oncology medical office, Herne
  - Marienkrankenhaus, Herne
  - Community based hemato-oncology medical office, Homberg (Ohm)
  - Community based hemato-oncology medical office, Kaiserslautern
  - Städtisches Klinikum, Karlsruhe
  - Community based hemato-oncology medical office, Kassel
  - Klinikum Kempten-Oberallgäu, Kempten
  - Community based hemato-oncology medical office, Koblenz
  - Community based hemato-oncology medical office, Krefeld
  - Community based hemato-oncology medical office, Kronach
  - Community based hemato-oncology medical office, Landau
  - Community based hemato-oncology medical office, Landshut
  - Klinikum Leverkusen GmbH, Leverkusen
  - St. Marienkrankenhaus, Ludwigshafen
  - Community based hemato-oncology medical office, Lüdenscheid
  - Universitätsklinik Mainz, Mainz
  - Community based hemato-oncology medical office, Marburg
  - Community based hemato-oncology medical office, Mönchengladbach
  - Community based hemato-oncology medical office, München
  - University Clinic Großhadern, München
  - Community based hemato-oncology medical office, Neumarkt
  - Community based hemato-oncology medical office, Nuremberg
  - St. Clemens Hospital, Oberhausen
  - St. Martinus-Hospital, Olpe
  - Community based hemato-oncology medical office, Osnabrück
  - St. Josefs-Krankenhaus, Potsdam
  - Community based hemato-oncology medical office, Rehling
  - Community based hemato-oncology medical office, Rüsselsheim am Main
  - Caritas Klinik St. Theresia, Saarbrücken
  - Community based hemato-oncology medical office, Schkeuditz
  - Kreiskrankenhaus Schotten, Schotten
  - Community based hemato-oncology medical office, Schweinfurt
  - Community based hemato-oncology medical office, Siegen
  - St.-Marien-Krankenhaus, Siegen
  - Diakonie - Klinikum Stuttgart, Stuttgart
  - Community based hemato-oncology medical office, Trier
  - Community based hemato-oncology medical office, Tübingen
  - University Clinic Ulm, Ulm
  - Städtisches Krankenhaus Villingen, Villingen-Schwenningen
  - Community based hemato-oncology medical office, Weilheim
  - Sophien- und Hufeland Klinikum, Weimar
  - Asklepios Nordseeklinik, Westerland
  - Community based hemato-oncology medical office, Wiesbaden
  - Dr. Horst-Schmidt-Kliniken, Wiesbaden
  - Community based hemato-oncology medical office, Wilhelmshaven
  - Community based hemato-oncology medical office, Wolfsburg

IPD SHARING:
Plan to Share IPD: No